CLINICAL TRIAL: NCT04076397
Title: Randomized Prospective Study Evaluating the Benefit of the Treatment of the Distal Amputation Sequelae of the Fingers by Lipofilling - LIPOFILLING Study
Brief Title: Lipofilling Versus Conservative Treatment in Fingertips Injuries Sequelae
Acronym: LIPOFILLING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC19.0081
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Distal Amputation of the Fingers
Keywords: annoying pulpal dysesthesia; lipofilling; amputation; sequelae
MeSH Terms: interventions — Desensitization, Psychologic

STUDY DESIGN:
Intervention Model Description: The randomization list is established by the Brest CHRU data management unit before the start of the trial. Based on a ratio (1: 1) with stratification on the center, the type of initial surgery (directed or flap scarring) and the duration of change of dysesthesia (≤ or> 1 year at baseline).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lipofilling group (Other): Patient will conduct a total of 4 visits: D15, M1, M3, M6 during which they will have: a clinical examination as well as the following evaluations:
  * Make EVA (evaluation of the pain),
  * Complete DASH questionnaire
  * Complete DN4 questionnaire
  Patients in the lipofilling group will also have:
  * the repair of the last dressing during the consultation at J15
  * Ablation of any threads
  * Control of the digital and abdominal scar
  * Making a photo of their finger at V1 and M6
  Interventions: Procedure: autologous transplant reinjection
- desensitization group (Other): Patient will conduct a total of 4 visits: D15, M1, M3, M6 during which they will have: a clinical examination as well as the following evaluations:
  * Make EVA (evaluation of the pain),
  * Complete DASH questionnaire
  * Complete DN4 questionnaire
  Interventions: Other: desensitization

INTERVENTIONS:
Procedure: autologous transplant reinjection — The patient is placed under loco-regional anesthesia. After sterilization of the upper limb and abdomen, the fat is removed at a fold by micro-incision by the Coleman method. The fat is decanted and micro-reinjected into the pulp of the patient's finger with 2 or 3 punctiform incisions. The quantity of fat injected is 2 to 3 mL. Incision of the abdomen and fingers is closed by points at monocryl 4/0. Finally, a fatty dressing is performed on the finger. Patients will benefit from nursing care every 2 days
  Arms: lipofilling group
Other: desensitization — Patients will have to stimulate the pulp of your finger on a daily basis
  Arms: desensitization group

SUMMARY:
The purpose of this study is to evaluate the contribution of autologous graft reinjection (lipofilling) in the treatment of dysaesthesic pulp.

ELIGIBILITY:
Inclusion Criteria:

* Major patient (18 years old) and ≤ 75 years old
* Patient with unidigital trauma downstream of distal interphalangeal joint
* Treated by directed healing OR covered by a flap
* Presenting troublesome pulpal dysesthesia evolving for more than 6 months AND less than 24 months
* The discomfort must be objectified by a DN4 score greater than or equal to 4/10 (neuropathic pain)
* Patient does not have any allergy to the substances used, in particular anesthetic: xylocaine, adrenaline

Exclusion Criteria:

* Patient with cutaneous sepsis, or amputation upstream of distal interphalangeal, or reimplantation, or dysesthesia that has been in progress for more than 24 months, or multi-digital traumatism
* Refusal of the patient to integrate the protocol Or incapacity to consent
* Pregnant or breastfeeding woman
* Tumor history of the amputated finger

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2028-04-02 (Estimated); Study Completion 2028-04-02 (Estimated)

PRIMARY OUTCOMES:
Decrease of the EVA between D0 and M6 | Day 0, Month 6
  visual analogue scale from 0 to 10, knowing that 0 is the absence of discomfort and intolerable discomfort

SECONDARY OUTCOMES:
Subjective self-assessment of the overall functional ability of both upper limbs | Day 0, Day 15, Month1, Month3, Month6
  DASH questionnaire (Disability of Arm-Shoulder-Hand)

OTHER OUTCOMES:
Neuropathic pain | Day 0, Day 15, Month 1, Month 3, Month 6
  DN4 score (questionnaire) : a score greater than or equal to 4 makes the diagnosis of neuropathic pain.
Patient satisfaction on the esthetic aspect of the finger | Month 6
  Subjective satisfaction to the patient's appreciation.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - CH de Cornouaille - Quimper, Quimper

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.